CLINICAL TRIAL: NCT01893918
Title: Assessment of Severity and Prognosis in Elderly Patients With Chronic Obstructive Pulmonary Disease (COPD) and Complex Chronic Comorbidities
Brief Title: Assessment of Severity and Prognosis in Elderly Patients With COPD and Complex Chronic Comorbidities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Leonardo M. Fabbri, Professor, University of Modena and Reggio Emilia
Other Study IDs: CCM147/10
Record Dates: First submitted 2013-02-01; First posted 2013-07-09 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: COPD
Keywords: Smoking; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Blood sampling for complete blood count, fasting glucose, bilirubin, creatinine, blood urea, uric acid, electrolytes (magnesium, sodium, potassium, chloride), total cholesterol, cholesterol high-density lipoprotein (HDL), triglycerides, serum glutamic oxaloacetic transaminase, serum glutamic pyruvic transaminase, gamma-glutamyl transpeptidase, creatine phosphokinase, hemoglobin A1c, serum insulin. Urine sampling for microalbuminuria and urine creatinine. Measurement of arterial blood gas. Blood sampling for biomarkers (NT-proBNP, high-sensitive C-Reactive Protein, IL-1β, IL-6).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- COPD patients: COPD patients, males and females, older than 65 years, with smoking history > 20 pack/years

SUMMARY:
Cigarette smoking, the major risk factor for Chronic Obstructive Pulmonary Disease (COPD), causes systemic effects, such as systemic cellular and humoral inflammation, that could substantially contribute to the development of chronic diseases, other than COPD, mainly cardiovascular diseases and metabolic disorders. Such chronic comorbidities affect health outcomes in COPD, particularly in terms of disease severity and prognosis. The aim of the project is to investigate the prevalence of chronic comorbidities associated with COPD and their impact on prognosis in elderly patients.

DETAILED DESCRIPTION:
The investigators will recruit 100 outpatients, heavy smokers (20 pack/years), older than 65 years, diagnosed with COPD. COPD is defined by presence of fixed airflow limitation: post-bronchodilator forced expiratory volume at one second (FEV1)/forced vital capacity (FVC) less than 70% according to spirometry classification from Global Inititiative for Obstructive Lung Disease (GOLD) guidelines. Each patient will be characterized by medical history, physical examination, and smoking history. Each patient will perform pulmonary function test, including reversibility to inhaled bronchodilator (400 mcg albuterol), and 6-minute walk test. Arterial blood gases and routine blood test, including inflammatory biomarkers, will also examined. In addition, each patient will undergo chest X-ray, thorax CT scan, echocardiography, and carotid ultrasonography.

At enrollment, all patients will be in stable condition (no changes in medication dosage or frequency, no COPD exacerbation or hospital admissions in the previous 4 weeks). Clinical and biological follow-up will be prospectively followed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians
* Age > 65 years
* Smoking history > 20 pack/years (current or former smokers)
* Diagnosis of COPD according to GOLD 2010
* Stable condition

Exclusion Criteria:

* History of bronchial asthma
* Other chronic diseases such as interstitial lung disease, bronchiectasis, bronchiolitis obliterans organizing pneumonia (BOOP), pulmonary tuberculosis, cystic fibrosis
* Malignancies for which patient is being treated with radiotherapy or chemotherapy
* Acute events and/or hospitalization within 12 weeks prior to screening

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 100 patients older than 65 years with diagnosis of COPD, current smokers or ex-smokers with more than 20 pack/years, in stable condition.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Number of chronic comorbidities associated to COPD | 0-3 years
  Number of comorbidities for the formulation of a severity score with predictive value to 3 years in terms of hospital admissions for acute events and mortality.

SECONDARY OUTCOMES:
Formulation of a severity score | 0-3 years
  A severity score will be developed on the basis of lung function impairment, different clinical phenotypes (chronic bronchitis and/or emphysema), and systemic inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo M Fabbri, MD, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- Azienda Ospedaliero-Universitaria di Modena, Modena, Italy